CLINICAL TRIAL: NCT05696106
Title: Risk of Incident Immune-mediated Inflammatory Diseases (IMID) in Patients Treated With Biologics and Immunosuppressive Drugs for a Single IMID
Brief Title: Risk of Incident IMID in Patients Treated With Biologics and Immunosuppressive Drugs for a Single IMID
Acronym: PROTECT-IMID
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC-21-0113
Record Dates: First submitted 2023-01-03; First posted 2023-01-25 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Inflammatory Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients initiating a biologic or immunosuppressive drug: Patients initiating a biologic or immunosuppressive drug including small molecules for a first IMID (either IBD, inflammatory rheumatic diseases, or cutaneous psoriasis)
  * Conventional immunosuppressive drug including immunomodulators (thiopurines) and csDMARDs (methotrexate)
  * Anti-TNF (infliximab, adalimumab, golimumab, certolizumab, etanercept)
  * Biologics targeting the IL-12/IL-23 pathways (ustekinumab, risankizumab, guselkumab)
  * Biologics targeting the IL-6 pathways (tocilizumab, sarilumab)
  * Biologics targeting the IL-17 pathways (secukinumab, ixékizumab, brodalumab)
  * Biologics targeting cell adhesion, anti-integrins (vedolizumab)
  * JAK inhibitors (tofacitinib, baricitinib, upadacitinib)

SUMMARY:
Individuals with immune-mediated inflammatory diseases (IMIDs) are at increased risk of developing other IMIDs, possibly through shared pathogenic inflammatory pathways, and up to 25% of patients with IMIDs have at least one other IMID. Additionally, a concomitant diagnosis of a second IMID is associated with a higher burden of disease, which usually requires therapeutic escalation. Thus, this risk should be taken into account in the benefit-risk balance of IMIDs-related treatment. While the risk of other major adverse events, such as serious infection, cancer, and cardiovascular events, have been assessed in patients exposed to immunosuppressive drugs and biologics, the impact of these drugs on the risk of incident IMIDs remains largely unknown.

The main aim of this study is to assess the risk of an incident second IMID in patients starting biologics including anti-TNF and immunosuppressive drugs including small molecules for a first IMID (either inflammatory bowel disease, inflammatory rheumatic diseases, or cutaneous psoriasis).

DETAILED DESCRIPTION:
This is a retrospective cohort study including all patients identified with a first IMID between 2008 and 2020 based on the French administrative healthcare databases (Système National des Données de Santé). Index date will be the date of initiation of the first treatment of interest within the observation period.

Primary objective

- To assess the risk of an incident second IMID in patients starting biologics including anti-TNF and immunosuppressive drugs including small molecules for a first IMID (either IBD, inflammatory rheumatic diseases, or cutaneous psoriasis)

Secondary objectives

* To describe the subtype of incident second IMIDs in patients starting biologics and immunosuppressive drugs for a first IMID and the related burden of disease.
* To assess the risk of an incident second IMID in patients starting biologics and immunosuppressive drugs for a first IMID, according to each drug class:

  * Conventional immunosuppressive drug including immunomodulators (thiopurines) and csDMARDs (methotrexate)
  * Anti-TNF (infliximab, adalimumab, golimumab, certolizumab, etanercept)
  * Biologics targeting the IL-12/IL-23 pathways (ustekinumab, risankizumab, guselkumab)
  * Biologics targeting the IL-6 pathways (tocilizumab, sarilumab)
  * Biologics targeting the IL-17 pathways (secukinumab, ixékizumab, brodalumab)
  * Biologics targeting cell adhesion, anti-integrins (vedolizumab)
  * JAK inhibitors (tofacitinib, baricitinib, upadacitinib)
* To assess the risk of an incident second IMID in patients with a first incident IMID (after January 1st, 2008) and starting biologics and immunosuppressive drugs for this IMID.
* To assess the risk of an incident second IMID in patients starting biologics and immunosuppressive drugs for a first IMID:

  * By type of first IMID
  * By type of second IMID

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older at index date (≥ 18 years)
* Identified with a first IMID diagnosis prior to index date, among IBD (Crohn's disease and ulcerative colitis), inflammatory rheumatic diseases (rheumatoid arthritis, ankylosing spondylitis, and psoriatic arthritis), or inflammatory skin diseases (psoriasis).

Exclusion Criteria:

* Patients with a diagnosis of more than one of the IMIDs of interest at index date.
* Patients exposed to biologics or immunosuppressive drugs of interest in 2006 or 2007.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the individual subtypes of second IMIDs included in the primary outcome definition, for which incidence during follow-up will be sufficient.
Sampling Method: Non-Probability Sample
Enrollment: 750000 (Estimated)
Dates: Start 2023-04-02 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of incident second IMID | between 1st January, 2008 and December 31st, 2018
  The primary outcome will be defined as the first occurrence of incident IMIDs after cohort entry, including: (Crohn's disease and ulcerative colitis, rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, psoriasis, systemic lupus erythematosus, drug-induced lupus, sarcoidosis, vasculitis, crohn's disease and ulcerative colitis, rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, psoriasis, systemic lupus erythematosus, drug-induced lupus, sarcoidosis, vasculitis). Identification algorithms used for inclusion criteria will be similarly used to assess outcomes. We performed a feasibility analysis by assessing the identification method of IBD diagnosis in patients previously diagnosed with either rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, or psoriasis. This analysis was based on a cohort of patients diagnosed with IBD between 1st January, 2008 and December 31st, 2018

SECONDARY OUTCOMES:
All the individual subtypes of second IMIDs included in the primary outcome definition | between 1st January, 2008 and December 31st, 2018
  All the individual subtypes of second IMIDs included in the primary outcome definition, for which incidence during follow-up will be sufficient.
  Burden of disease will be based on healthcare resource utilization, notably hospitalizations, emergency department visits, outpatient visits, and drug deliveries.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint-Antoine, Paris, France